Study Number: UX023-CL203 Statistical Analysis Plan Amendment 1

27 April 2016, Version 1.1



#### STATISTICAL ANALYSIS PLAN

Title A Phase 2b, Open-Label, Long-Term Extension Study

to Evaluate the Safety and Pharmacodynamics of

KRN23 in Adult Subjects with X-Linked

Hypophosphatemia (XLH)

**Protocol:** UX023-CL203

Investigational Product: KRN23 (Recombinant human IgG1 monoclonal

antibody to fibroblast growth factor 23 [FGF23])

**Indication:** X-linked Hypophosphatemia (XLH)

IND/EudraCT Number: 076488

PPD **Author:** 

Consultant, Biostatistics

Ultragenyx Pharmaceutical Inc.

60 Leveroni Court

Novato, CA, USA 94949

Date: 27 April 2016

**Version Number:** 1.1



## STATISTICAL ANALYSIS PLAN AMENDMENT

#### **SUMMARY OF CHANGES**

#### UX023-CL203 Amendment 1

## 27 April 2016

The UX023-CL203 statistical analysis plan (dated 15 January 2016) has been amended. Important changes in Amendment 1 are summarized below:

- 1. **Interim Analysis Timing**: Section 3.6 has been updated to reflect the timing of the interim analysis to support regulatory submission.
- **2.** Events to Monitor: Section 8.6.1 has been updated so that the events to monitor categories are consistent with the product identified or potential risks.
- **3. Analysis of Vital Signs**: Section 8.6.6 has been updated to reflect the standard descriptive analysis for vital signs.
- **4. Analysis of ECG**: Section 8.7.2 has been updated to remove the normality or abnormality analysis of the ECG tracing because the overall interpretation of ECG is not collected for the study.
- **5. 6-Minute Walk Test**: Section 8.8.2.3 has been updated to remove the graph display of 6-minute walk test data because there is only one post-baseline time point (Week 24).



# **Table of Contents**

| 1 | INT | RODUCTION | 8 |
|---|---|---|---|
| 2 | STU | JDY OBJECTIVES | 9 |
| | 2.1 | Primary Safety and Pharmacodynamics | 9 |
| | 2.2 | Efficacy | 9 |
| 3 | STU | JDY DESIGN | 10 |
| | 3.1 | Overall Study Design and Plan | 10 |
| | 3.2 | Study Duration | 10 |
| | 3.3 | Randomization and Blinding Method of Assigning Subjects to Treatment Groups | 10 |
| | 3.4 | Stratification Factors | 10 |
| | 3.5 | Determination of Sample Size | 11 |
| | 3.6 | Week 24 Analysis | 11 |
| | 3.7 | Data Monitoring Committee | 11 |
| 4 | STU | DY CLINICAL OUTCOMES AND COVARIATES | 12 |
| | 4.1 | Safety Endpoints | 12 |
| | 4.2 | Pharmacodynamics Endpoints | 12 |
| | 4.3 | Efficacy Endpoints | 12 |
| 5 | DEF | FINITIONS AND DERIVED EFFICACY VARIABLES | 13 |
| | 5.1 | Baseline | 13 |
| | 5.2 | First KRN23 Dose Date | 13 |
| | 5.3 | BPI | 13 |
| | 5.4 | WOMAC | 13 |
| | | 5.4.1. MPCI for WOMAC Scales and Responder definition | 14 |
| | 5.5 | SF-36 Health Survey version 2 | 15 |
| | | 5.5.1 MIC for SF-36v2 Scales and Responder definition | 16 |
| | 5.6 | Percent of Predicted 6-Minute Walk Test Distance | 17 |
| | 5.7 | Events To Monitor | 17 |



| 6 | ANA | ALYSIS | POPULATIONS | 18 |
|---|---|---|---|---|
| | 6.1 | Safety | Analysis Set | 18 |
| | 6.2 | Pharma | acodynamic Analysis Set | 18 |
| | 6.3 | Efficac | cy Analysis Set | 18 |
| 7 | DA | ΓA SCR | EENING AND ACCEPTANCE | 19 |
| | 7.1 | Handli | ng of Missing and Incomplete Data | 19 |
| | 7.2 | Missin | g data in WOMAC questionnaire | 19 |
| | 7.3 | Missin | g data in SF36 questionnaire | 19 |
| | 7.4 | Missin | g Date Imputation Rules. | 19 |
| | 7.5 | Unsche | eduled or Early Termination Visits | 20 |
| | 7.6 | Softwa | nre | 20 |
| 8 | STA | TISTIC | AL METHODS OF ANALYSIS | 21 |
| | 8.1 | Genera | al Principles | 21 |
| | | 8.1.1 | Repeated Measure Model: General Estimating Equations | 21 |
| | | 8.1.2 | Graphic Displays and Study Results | 22 |
| | | 8.1.3 | Direction of Effects for the PRO Endpoints | 22 |
| | 8.2 | Demog | graphics and Baseline Characteristics | 22 |
| | 8.3 | Diseas | e Characteristics and Medical History | 22 |
| | | 8.3.1 | Medical History / XLH Medical History | 22 |
| | | 8.3.2 | XLH Treatment History | 22 |
| | 8.4 | Subjec | t Accountability | 22 |
| | 8.5 | Dosing | g Summary | 23 |
| | 8.6 | Genera | al Safety | 23 |
| | | 8.6.1 | Adverse Events | 23 |
| | | 8.6.2 | Safety Lab Parameters | 24 |
| | | 8.6.3 | Concomitant Medications | 24 |
| | | 8.6.4 | Physical Examination | 24 |



| | | 8.6.5 | Pregnand | cy Test | 24 |
|---|---|---|---|---|---|
| | | 8.6.6 | Vital Sig | gns | 25 |
| | 8.7 | Ectopi | ic Mineraliz | zation Safety | 25 |
| | | 8.7.1 | Renal U | ltrasound | 25 |
| | | 8.7.2 | ECG | | 25 |
| | | 8.7.3 | ЕСНО | | 25 |
| | 8.8 | Endpo | oints | | 26 |
| | | 8.8.1 | Pharmac | odynamic Endpoints | 26 |
| | | 8.8.2 | Efficacy | Endpoints | 26 |
| | | | 8.8.2.1 | PRO Endpoints | 26 |
| | | | 8.8.2.2 | X-Ray Endpoints | 27 |
| | | | 8.8.2.3 | 6-Minute Walk Test and Percent Predicted 6-Minute Walk Test | 27 |
| | | | 8.8.2.4 | Timed Up and Go Test | 27 |
| | | | 8.8.2.5 | Subgroup Analyses | 27 |
| 9 | REF | EREN | CES | | 28 |
| 10 | APP | ENDIC | EES | | 29 |
| | App | endix 1 | : UX023-C | L203 Efficacy Endpoint Summary Table | 29 |
| | App | endix 2 | : BPI Ques | tionnaire | 33 |
| | App | endix 3 | : WOMAC | Questionnaire | 35 |
| | App | endix 4 | : SF-36 Qu | estionnaire | 38 |
| | App | endix 5 | : Events to | Monitor | 44 |
| | App | endix 6 | : Schedule | of Events | 56 |



# **List of Tables**

| Table 1: WOMAC Scales, Number of Questions in Each Scale, and Scores from a | |
|---|---|
| General Population. | 14 |
| Table 2: SF-36v2 Scales and Number of Questions in Each Scale | 15 |
| List of Figures | |
| Figure 1: Process for scoring SF-36v2 Health Domain Scales and Component | |
| Summary Measures | 1 <i>6</i> |

Study Number: UX023-CL203 Statistical Analysis Plan Amendment 1

27 April 2016, Version 1.1



#### **ABBREVIATIONS**

1,25[OH]<sub>2</sub>D 1,25-dihydroxyvitamin D 3MSCT 3-Minute Stair Climb Test

6MWT 6-Minute Walk Test

AE Adverse event

ALP Alkaline phosphatase

BALP Bone-specific alkaline phosphatase

BMI Body mass index
BPI Brief Pain Inventory
CFB Change from Baseline

CTx Carboxy terminal cross-linked telopeptide of type I collagen

FGFR1 Fibroblast growth factor receptor 1

FGF23 Fibroblast growth factor 23

GEE Generalized Estimating Equations

GFR Glomerular filtration rate
HAHA Anti-KRN23 antibody
HQRL Health-related quality of life
iPTH Intact parathyroid hormone
ISR Injection site reactions
LVH Left ventricular hypertrophy

mAb Monoclonal antibody

MedDRA Medical Dictionary for Regulatory Activities P1NP Procollagen type 1 N-terminal propeptide

PD Pharmacodynamic

PHEX Phosphate-regulating gene with Homologies to Endopeptidases on the X-

chromosome

PRO Subject-reported outcome

QOL Quality of life

QTc Corrected QT interval SAE Serious adverse event

SC Subcutaneous

SF-36 36-item Short Form Health Survey SMQ Standardised MedDRA Query TEAE Treatment-emergent adverse event

TmP/GFR Ratio of renal tubular maximum phosphate reabsorption rate to glomerular

filtration rate

TRP Tubular resorption of phosphate

TUG Timed up and go

WHO World Health Organization

WOMAC Western Ontario and McMaster Universities Osteoarthritis Index

XLH X-Linked Hypophosphatemia



## 1 INTRODUCTION

The purpose of this statistical analysis plan is to provide details of the statistical analyses that have been outlined within the original UX023-CL203 Protocol dated 05 September 2014. The data collected in this study will evaluate the safety and pharmacodynamics of KRN23 in adult subjects with X-Linked Hypophosphatemia.



#### 2 STUDY OBJECTIVES

## 2.1 Primary Safety and Pharmacodynamics

The primary objectives of this study are to:

- Assess the long-term safety of KRN23 SC administration in adult subjects with XLH
- Assess the proportion of subjects achieving serum phosphorus levels in the normal range (2.5-4.5 mg/dL) with long-term administration of KRN23
- Assess long-term PD of KRN23 as measured by changes in the following:
  - Serum and urinary phosphorus
  - TmP/GFR and TRP
  - Serum 1,25(OH)<sub>2</sub>D
  - Serum FGF23
  - Bone biomarkers: serum ALP, bone-specific ALP (BALP), carboxy terminal crosslinked telopeptide of type I collagen (CTx), and procollagen type 1 N-terminal propeptide (P1NP)
- Assess long-term immunogenicity of KRN23 as measured by presence of anti-KRN23 antibody (HaHa)

#### 2.2 Efficacy

The efficacy objectives of this study are to:

- Evaluate changes in underlying skeletal disease by standard radiographs of the legs, feet, and lateral spine as well as any location(s) where the subject is currently experiencing tenderness or pain that may reflect underlying pathology, or where the subject has a history of recent (< 3 months) fracture
- Evaluate changes in subject-reported outcomes (PROs) and physical function outcomes including:
  - Subject-reported pain Brief Pain Inventory (BPI)
  - Disability Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
  - Quality of life (QOL) scores 36-item Short Form Health Survey (SF-36)
  - Walking ability 6-Minute Walk Test (6MWT)
  - Balance and agility Timed Up and Go (TUG) Test

Due to the inability to standardize the number of stairs used for testing at all study sites, the 3MSCT was not collected in this study and is excluded from the final and interim analyses.



## 3 STUDY DESIGN

## 3.1 Overall Study Design and Plan

This study is a Phase 2b, open-label, long-term extension study of the completed studies KRN23-INT-001 and KRN23-INT-002 in adult subjects with XLH. The study population will consist of approximately 25 eligible subjects who participated in Kyowa Hakko Kirin Pharma, Incorporated's study KRN23-INT-001 or study KRN23-INT-002 (received at least 2 doses of KRN23). Subjects who were discontinued from KRN23-INT-001 or KRN23-INT-002 due to a TEAE classified as possibly or probably related to treatment may be eligible for participation in this study based on the clinical judgment of the investigator with agreement from the sponsor. The study will be conducted over 72 weeks to assess the long-term safety, immunogenicity, PD, and clinical efficacy of KRN23.

The starting dose of KRN23 at Baseline (Week 0) in this study will be individual for each subject, i.e., the same as a subject's last dose in studies KRN23-INT-001 or KRN23-INT-002 (0.30, 0.60, or 1.0 mg/kg). Dosing will occur at the clinic and the volume will be based on the weight obtained on Day 0.

Up to Week 12, individual subjects who have not reached serum phosphorus levels above the lower limit of normal (LLN; 2.5 mg/dL) at the end of the dose interval may have their doses titrated every 4 weeks to a maximum dose of 1.0 mg/kg based on fasting trough serum phosphorus levels. Doses may be titrated downward if at any point the serum phosphorus level increases above the upper limit of normal (ULN; 4.5 mg/dL). KRN23 injections will be repeated every 4 weeks for the duration of the study (from Week 0 through Week 68), and weight will be reassessed periodically for dose volume adjustments as needed.

A complete schedule of events is included in Appendix 6.

## 3.2 Study Duration

The planned duration of treatment in this study will be 72 weeks.

## 3.3 Randomization and Blinding Method of Assigning Subjects to Treatment Groups

All subjects received KRN23 on an open-label basis. Randomization and blinding are not applicable in this study.

#### 3.4 Stratification Factors

Not applicable.



## 3.5 Determination of Sample Size

The rationale for the sample size for this open-label extension study is based on practical considerations to obtain the needed information to meet study objectives. The sample size of this study is based on the number of subjects who have satisfactorily completed studies KRN23-INT-001 and/or KRN23-INT-002, along with the other eligibility criteria, and have agreed to participate in this long-term extension study. Approximately 25 subjects may be enrolled in this study. Subjects who were enrolled in the KRN23-INT-002 bone sub-study and who received KRN23 are also eligible. Since this is an exploratory study, no formal statistical power and sample size estimation methods were used to determine the sample size; therefore, the current study design is not powered to assess a pre-defined statistical difference in any endpoint.

## 3.6 Week 24 Analysis

Week 24 analysis will be conducted after all subjects have completed the Week 24 visits or discontinued the study. The purpose of this analysis is to potentially provide supporting data to any regulatory filings of UX023 in XLH.

Additional interim analyses may be conducted if deemed necessary.

## 3.7 Data Monitoring Committee

Based on the open-label study design, safety will be monitored by Ultragenyx. An independent data monitoring committee will not be used.



#### 4 STUDY CLINICAL OUTCOMES AND COVARIATES

## 4.1 Safety Endpoints

Safety assessments will be summarized at Baseline and at each observed time that they are collected. In addition to the incidence and frequency of AEs, the following endpoints will be examined as CFB:

- Number of clinically significant changes in vital signs, laboratory tests, physical examinations, ECHO and ECG, and renal ultrasounds
- Number of subjects who develop anti-KRN23 antibodies

## 4.2 Pharmacodynamics Endpoints

The primary pharmacodynamics endpoints are:

- Number and percentage of subjects who have serum phosphorus levels which, at any time after dosing are in the normal range ( $\geq 2.5$  and  $\leq 4.5$ ) or outside the normal range
- Change from baseline in serum biochemistry parameters associated with XLH, as measured by serum phosphorus, iPTH, FGF23 (total and free), and 1,25(OH)<sub>2</sub>D
- Change from baseline in urinalysis parameters associated with XLH, as measured by 2-hour urine TmP/GFR and TRP, i.e., calcium, creatinine, and phosphorus
- Change from baseline in urine parameters associated with XLH, as measured by 24-hour urine, i.e., urinary phosphate, calcium, creatinine, and urine calcium/creatinine ratio
- Change from baseline in bone biomarkers associated with XLH, as measured by total ALP and BALP, CTx, and P1NP
- Change from baseline in fractional excretion of phosphorus (FEP), defined as 100%\*(2-hour urine phosphorus\*serum creatinine)/(2-hour urine creatinine \* serum phosphorus)

## 4.3 Efficacy Endpoints

The exploratory efficacy endpoints are:

- Change from baseline in pain and health-related QoL as measured by changes in the WOMAC, BPI, and SF-36 scores
- Healing of prior or existing fractures or other disease-related skeletal abnormalities as viewed on standard radiographs
- Change from baseline in walking ability as measured by change in the distance walked on the 6MWT in meters and percent predicted normal values
- Change from baseline in transitions during ambulatory activity that incorporates strength, agility, and dynamic balance as measured by the time required to complete the TUG test.



#### 5 DEFINITIONS AND DERIVED EFFICACY VARIABLES

#### 5.1 Baseline

Baseline is defined as the last non-missing measurement taken prior to the first dose of study drug administration in CL203 study.

Note that all subjects enrolled in this study received at least 2 doses of KRN23 in Kyowa Hakko Kirin Pharma, Incorporated's study KRN23-INT-001 or study KRN23-INT-002; however, since a minimum of 21 months separated the last dose in KRN23-US-001/002 studies and the first dose in this study, values measured in KRN23-INT-001 or KRN-INT-002 studies will not serve as baseline values for this study.

## 5.2 First KRN23 Dose Date

First KRN23 dose date refers to the first dose of KRN23 given in UX023-CL203 study. First dose date will not take into account KRN23 doses given in studies KRN23-US-02, KRN23-INT-001 or KRN23-INT-002.

#### 5.3 **BPI**

The BPI will be completed by subjects to assess pain severity and the impact of pain on daily functioning.

The BPI endpoints to be analyzed are as follows:

- Worst pain, defined as the answer to question 3 (pain at its worst in the last 24 hours)
- Pain severity, defined as the average of questions 3 through 6
- Pain interference, defined as the average of questions 9A through 9G regarding "pain interfered" in the last 24 hours.

Appendix 2 includes the complete text of the BPI. Of note, subjects enrolled in this study were not asked questions 7 and 8, therefore the answers to these questions are not used for analysis in this study.

#### 5.4 WOMAC

The WOMAC will be completed by subjects to assess pain, stiffness, and physical function. The WOMAC consists of 24 items divided into 3 subscales:

- Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing
- Stiffness (2 items): after first waking and later in the day
- Physical Function (17 items): stair use, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in



bed, getting in / out of bath, sitting, getting on / off toilet, heavy household duties, light household duties.

The 24-question self-reported WOMAC evaluates the condition of the knee, hip, and other joints in osteoarthritis, measuring three dimensions: Pain, Stiffness, and Physical Functioning (Table 1) over the previous 48 hours.

Table 1: WOMAC Scales, Number of Questions in Each Scale, and Scores from a General Population

| | | Normative valu popul | es from general ation <sup>1</sup> |
|---|---|---|---|
| Scale Name | Number of WOMAC questions combined into scale score | Mean* | Standard<br>Deviation* |
| Pain | 5 | 14.1 | 19.7 |
| Stiffness | 2 | 20.1 | 23.6 |
| Physical Functioning | 17 | 15.4 | 20.2 |

<sup>\*</sup> The published values are on a 0-10 scale and were converted here to a 0-100 scale by multiplying by 10.

All questions are measured on a 5-point Likert scale: none (0), mild (1), moderate (2), severe (3), and extreme (4). Scoring is a simple sum, so Pain scores could range from 0 to 20, Stiffness from 0 to 8, and Physical Functioning from 0 to 68, with higher numbers indicating worse condition. Scores are then normalized to a 0-100 metric representing the percent of the maximum score, where 0 was the best health state and 100 the worst.

WOMAC scores are not norm-based, so they cannot be interpreted directly as difference from a population mean. However, mean WOMAC scores from a large population-based sample of healthy adults have been published (Bellamy et al. 2011), giving benchmark values for comparison (Table 1).

Appendix 3 includes the complete text of the WOMAC as it appears to subjects in the study.

## 5.4.1. MPCI for WOMAC Scales and Responder definition

The minimum perceptible clinical improvement (MPCI) for WOMAC scales are defined according to the WOMAC User Guide (Bellamy 2012) as follows:

- WOMAC Pain: 9.7 nu (normalized units)
- WOMAC Stiffness: 10.0 nu
- WOMAC Physical Functioning: 9.3 nu

For each of the three WOMAC scales the responders are the subjects with the decrease from baseline greater than or equal to the corresponding MPCI.



## 5.5 SF-36 Health Survey version 2

The SF-36v2 is a self-reported survey of general HRQL with a 4-week recall period. Its 36 questions measure eight underlying health domains, and responses to sets of questions are combined and scored to yield scale scores for each domain, as shown in Table 2.

Table 2: SF-36v2 Scales and Number of Questions in Each Scale

| Scale Name | Acronym | Number of SF-36v2 questions combined into scale score |
|---|---|---|
| Physical Functioning | PF | 10 |
| Role Limitations due to Physical Health | RP | 4 |
| Bodily Pain | BP | 2 |
| General Health Perceptions | GH | 5 |
| Vitality | VT | 4 |
| Social Functioning | SF | 2 |
| Role Limitations due to Emotional Problems | RE | 3 |
| Mental Health | МН | 5 |

Note: The health transition question (item 2 on the SF-36v2, as shown in Appendix 4) is not used in the calculation of SF-36v2 scales.

Additionally two summary component scores are calculated from domain scores (Physical Component Summary Scale [PCS] and the Mental Component Summary Scale [MCS]). They each draw information from all eight scales, with weights derived from the population-based sample. The PCS depends most heavily on the PF, RP, BP and GH scales, while the MCS mainly reflects the MH, RE, SF, and VT scales.

Raw scores range from 0 to 100 with higher scores indicating better health. Domain scores are calculated from raw scores such that domain scores have a mean of 50 and SD of 10. The PCS and MCS summary component scores also have mean of 50 and SD of 10 to allow comparisons with domain scores.

Scoring the SF-36 version 2 is accomplished using T-score Based scoring software from QualityMetric Inc (Maruish 2011). T-score Based scoring is standardized across the SF family of adult tools using the means and standard deviations from the 2009 U.S. general population. The T-score Based scores in the U.S. general population have a mean of 50 and a standard deviation of 10. The PCS and MCS are both expressed as norm-based scores on the



same metric as the scales, and can be interpreted in the same manner. The scoring process is summarized in Figure 1.

The main advantage of T-score Based scoring of the adult SF tools is easier interpretation. By using the T-score Based scoring method, the data are scored in relation to U.S. general population t-scores. Therefore, all scores obtained that are below 40 can be interpreted as 1 standard deviation below the U.S. general population t-score and scores above 60 can be interpreted as 1 standard deviation above the U.S. general population t-score. Because the standard deviation for each scale is 10, it is easier to see exactly how far above or below the mean a score is in standard deviation units (10 points = 1 standard deviation unit).

Appendix 4 includes the complete text of the SF-36 as it appears to subjects in the study.

Figure 1: Process for scoring SF-36v2 Health Domain Scales and Component Summary Measures



## 5.5.1 MIC for SF-36v2 Scales and Responder definition

The Minimally Important Change (MIC) is the smallest change over time in an individual patient's score that represents a clinically significant change in their health status. Using a distributional approach with a US general population sample, MICs have been established for the SF-36v2 as: PF, 3.5 points; Role-Physical, 3.2; Bodily Pain, 4.5; General Health, 5.7; Vitality, 5.5; Social Functioning, 5.0; Role-Emotional, 3.8; Mental Health, 5.5; PCS, 3.1; and MCS, 3.8.



## 5.6 Percent of Predicted 6-Minute Walk Test Distance

To calculate the percent predicted 6MWT value, the following formula will be applied (Gibbons et al. 2001).

$$X_i = \frac{X_{0i}}{868.8 - (2.99 \times Age) - (74.7 \times Gender)} * 100$$

where  $X_i$  is the percent predicted 6MWT result at time i for subject X,  $X_{0i}$  is the 6MWT result (in meters) at time i for subject X, and Gender is equal to 0 if the subject is male or 1 if the subject is female. Age at the study visit will be used for the calculation for the duration of the study.

#### 5.7 Events To Monitor

**Injection Site Reaction (ISR)**: Defined by preferred terms under the Medical Dictionary for Regulatory Activities (MedDRA) high-level term (HLT) "Injection site reaction".

**Immunogenicity AE**: Defined using relevant PTs in the narrow SMQs for "Hypersensitivity".

**Hyperphosphataemia AE**: Defined by using PTs: "Hyperphosphataemia", "Blood phosphorus increased".

**Ectopic calcification related AE**: There is no available SMQ. Ectopic calcification related AE is defined using a MedDRA search of 'calcification'.

**Gastrointestinal AEs:** i.e. nausea, vomiting, abdominal pain, diarrhea. Defined using PTs in the narrow SMQ "Gastrointestinal nonspecific inflammation and dysfunctional conditions".

**Restless leg syndrome AE**:. Defined by PTs "Restless legs syndrome", "Restlessness", "Akathisia", "Sensory disturbance", "Psychomotor hyperactivity", "Limb discomfort", "Neuromuscular pain", "Formication".

See search criteria in Appendix 5.



## **6 ANALYSIS POPULATIONS**

## 6.1 Safety Analysis Set

The safety analysis population will consist of all enrolled subjects who receive at least 1 dose of KRN23 (full or partial injection) during the study.

## 6.2 Pharmacodynamic Analysis Set

The pharmacodynamic (PD) analysis set consists of all subjects who receive at least 1 dose of study drug and who have evaluable plasma/serum data.

## 6.3 Efficacy Analysis Set

All efficacy analyses (other than the PD analyses) will be performed on all subjects who receive at least 1 dose of study drug and who have at least one pre- and post-treatment measurement.



#### 7 DATA SCREENING AND ACCEPTANCE

## 7.1 Handling of Missing and Incomplete Data

Missing clinical outcome data can occur for multiple reasons, including missed subject visits and scales or measures with missing item scores. Missing and incomplete data will be identified through a review of tables and listings for this study. Missing and incomplete data will be identified for investigation, and possible resolution, by Data Management prior to the study database lock.

For all analyses, missing data will be treated as missing, unless otherwise specified. When a change from baseline is assessed, only subjects with a baseline and at least one post-baseline measurement will be included in the analysis.

Depending on the number of discontinuations and missed visits from the study, a sensitivity analysis might be conducted for the pharmacodynamics and the efficacy endpoints analyses, where missing data will be imputed using mBOCF (modified Baseline Observation Carried Forward) defined as follows:

- for discontinuations due to AE or death use the worst between BOCF (Baseline Observation Carried Forward) and LOCF (Last Observation Carried Forward)
- otherwise use LOCF.

# 7.2 Missing data in WOMAC questionnaire

For computing the domain scores at each visit for each subject, the WOMAC missing data algorithm is as follows:

- 1. If two or more Pain items, both Stiffness items, or four or more Physical Functioning items are missing, then the corresponding scale score is set to missing.
- 2. Otherwise, any missing item is replaced with the mean of the other items in its scale, and scales are then calculated normally.

#### 7.3 Missing data in SF36 questionnaire

The SF-36v2 missing data algorithm for computing the domain scores from responses to individual items is property of QualityMetric, and is not available for further description.

## 7.4 Missing Date Imputation Rules

The following conventions will be used to impute missing portions of dates for adverse events and concomitant medications. Note that the imputed values outlined here may not always provide the most conservative date. In those circumstances, the imputed value may be replaced by a date that will lead to a more conservative analysis.

#### 1. Start Dates



- 1. If the year is unknown, then the date will not be imputed and will be assigned a missing value.
- 2. If the month is unknown, then:
  - 1. If the year matches the first dose date year, then impute the month and day of the first dose date.
  - 2. Otherwise, assign 'January.'
- 3. If the day is unknown, then:
  - 1. If the month and year match the first dose date month and year, then impute the day of the first dose date.
  - 2. Otherwise, assign the first day of the month.

## 2. Stop Dates

- 1. If the year is unknown, then the date will not be imputed and will be assigned a missing value.
- 2. If the month is unknown, then assign 'December.'
- 3. If the day is unknown, then assign the last day of the month.

## 7.5 Unscheduled or Early Termination Visits

In general, data collected by study visit will be summarized using the visit number specified in the database. Outcomes scheduled at a planned study visit but are collected during an unscheduled visit or early termination visit will be mapped into the closest study visit based on the study day of the unscheduled visit or early termination visit, and the schedule of assessment in the protocol.

For outcomes where both the planned study visit and an unscheduled visit or early termination visit corresponding to that study visit are both available, the planned study visit measurement will be used for the analysis.

All safety data including the planned study visits and unscheduled/early termination visits will be included in the shift tables.

All data will be included in the data listings and outcomes measured during unscheduled visits and early termination visits will be marked as acquired during an unscheduled visit.

#### 7.6 Software

SAS® software version 9.4 or higher will be used to perform most or all statistical analyses.



#### 8 STATISTICAL METHODS OF ANALYSIS

## 8.1 General Principles

The statistical analyses will be reported using summary tables, figures, and data listings. Statistical tests will be 2-sided at the alpha=0.05 significance level and 2-sided 95% confidence interval will be used. All p-values will be presented as nominal p-values. No adjustment on multiplicity will be made. Continuous variables will be summarized with means, standard deviations, standard errors, medians, Q1, Q3, minimums, and maximums. Categorical variables will be summarized by counts and by percentages of subjects in corresponding categories. No imputation on missing data will be made, unless stated otherwise. All data obtained from the CRFs as well as any derived data will be included in data listings.

The Week 24 analysis will be performed when all patients enrolled in the study have completed the Week 24 visit or have discontinued the study. The final analysis will be conducted when all patients enrolled in the study have completed the Week 72 visit or have discontinued the study.

# **8.1.1** Repeated Measure Model: General Estimating Equations

When the sample size and number of observations allow it, the change from baseline over time and the binary endpoints over time will be analyzed using a generalized estimation equation (GEE) model that includes time as the categorical variable and adjusted for baseline measurement. The covariance structure that will be used for the GEE model is compound symmetry which specifies constant variance for the assessments and constant covariance between the assessments over time. If the compound symmetry covariance structure leads to non-convergence, Quasi-Likelihood Information Criterion (QIC) will be used to select the best covariance structure. Model based estimates of the changes from baseline and corresponding 95% confidence intervals will also be provided along with p-values for assessing statistical significance.

The p-value for testing the statistical significance of the change from the baseline to week 24 (for the interim analysis) and to week 72 (for the final analysis) assessments will be provided for changes from baseline in primary PD endpoints, selected safety endpoints (eGFR, creatinine, amylase), PRO endpoints (BPI, WOMAC, SF-36) and clinical outcomes endpoints (6MWT, percent predicted 6MWT, TUG).

For week 24 analysis, only measurements up to week 24 will be included in the model. For final analysis (week 72), all measurements will be included in the model.

If the number of observations are insufficient for analyses using a GEE model, a descriptive summary will be provided, and analyses using observations at a single time point, such as paired t-test or nonparametric methodologies, will be considered.



## 8.1.2 Graphic Displays and Study Results

Graphical displays of study endpoints will be completed and include both observed study data and modeled analyses, where applicable. Arithmetic means, least square means (where applicable), and appropriate measure of dispersion (e.g., standard deviation, standard error) or confidence intervals may be displayed in figures. In general, graphical displays will accompany each planned analysis to present study results.

## 8.1.3 Direction of Effects for the PRO Endpoints

The three PRO endpoints for the study are not scaled in the same directions. In the SF-36v2 a higher score indicated better health whereas in the BPI and WOMAC higher scores indicate worse health. They are presented as-is, with reminders that improvements in health appear as positive numbers for the SF-36v2 and BPI scales and as negative numbers for the WOMAC scales.

## 8.2 Demographics and Baseline Characteristics

Summaries of demographic characteristics will include descriptive statistics for age, height, weight, BMI, renal ultrasound scores, baseline skeletal survey radiographs measures (mean, standard deviation, median, minimum and maximum values) and for sex, race, ethnicity, PHEX mutation, radiograph location (number and percentage of subjects in each category).

#### 8.3 Disease Characteristics and Medical History

## 8.3.1 Medical History / XLH Medical History

Medical history will be summarized by body system and will also be listed by subject.

#### **8.3.2** XLH Treatment History

A summary of subjects' past XLH treatment with oral phosphate (e.g., K-Phos, Phospha, Phosphate-Sandoz) and vitamin D metabolite (e.g. Calcitriol, Rocaltrol, alfacalcidol, Alpha-calcidol/1,alpha, 1,25 Vitamin D3, dihydrotachysterol) therapy will be presented. Use of calcimimetics or the treatment of hyperparathyroidism will also be reported. For subjects receiving standard of care therapy for XLH (phosphate and/or vitamin D) the drug name, duration of treatment, dose and frequency of administration will be listed. A summary of currently used walking devices will be included.

#### 8.4 Subject Accountability

Subject disposition summaries will include the number of subjects who received study medication, the number of subjects who completing the study, and the reasons for study discontinuation. The number of subjects included in the safety, pharmacodynamics and efficacy analysis, respectively, will be presented.



## 8.5 Dosing Summary

The total dose administered, weight-based dose will be summarized by study visit for the Safety Population. Study medication dispensing and treatment compliance will be summarized in individual subject listings.

## 8.6 General Safety

All safety analyses will be performed on the safety analysis set, unless stated otherwise. General safety will include AEs, treatment related AEs, SAEs, AE of injection site reaction (grouped by High-Level Group Term), laboratory measurements including chemistry, hematology, and urinalysis parameters, GFR, amylase, HAHA, concomitant medications, physical exams, pregnancy test and vital signs. No hypothesis testing is planned for safety data.

#### **8.6.1** Adverse Events

Reported adverse event (AE) terms are coded to MedDRA (version 18.1). All reported events will appear in AE listings, however only TEAE will be summarized. TEAEs are defined as AEs with onset on or after the time of initiation of study drug administration.

The following AEs will be summarized:

- All TEAEs
- Related TEAEs
- Events to monitor:
  - Injection site reactions
  - Gastrointestinal events
  - Immunogenicity
  - Ectopic mineralization
  - Hyperphosphatemia
  - Restless legs syndrome
- Grade 3/4 TEAEs
- Serious TEAEs
- Serious related TEAEs
- TEAEs resulting in discontinuation
- Fatal TEAEs.

Summaries of TEAEs will show incidence rates for each MedDRA primary SOC and PT.



All TEAEs will be tabulated in the following manner: by system organ class/preferred term in descending order, by system organ class/preferred term/relationship to study drug, and by system organ class/preferred term/severity. Additionally, treatment-emergent SAEs and TEAEs related to investigational drug will be tabulated by system organ class/preferred term in descending order.

Injection site reactions (ISR) will be listed for PT, seriousness, severity, outcome, relationship to study drug, and onset time from investigational product administration.

# 8.6.2 Safety Lab Parameters

The descriptive statistics will be provided for lab safety parameters (chemistry, hematology, and urinalysis parameters, GFR, HAHA). In addition, shift tables will be provided for HAHA (with categories Yes/No) and for amylase. For amylase, the following categories will be used:

- Normal
- Grade 1: 1 1.5 x ULR
- Grade 2: 1.5 2 x ULR
- Grade 3: 2 5 x ULR
- Grade 4:  $> 5 \times ULR$ .

#### **8.6.3** Concomitant Medications

Each medication will be coded to a preferred name and an Anatomic Therapeutic Classification (ATC) code using WHODrug. The number and percentage of subjects taking each concomitant medication will be displayed by preferred name. This display will be created for the safety analysis set. A concomitant medication listing will also be made. Prior medications, i.e. medications that were used within 30 days before the Screening visit will also be listed.

## 8.6.4 Physical Examination

Physical exam results will include the assessment of general appearance; head, eyes, ears, nose, and throat (HEENT); the cardiovascular, dermatology, lymphatic, respiratory, gastrointestinal, musculoskeletal, genitourinary, neurological systems All physical examination assessments will be listed.

#### 8.6.5 Pregnancy Test

Subject level listing for pregnancy test results will be created for those who had positive pregnancy test.



## 8.6.6 Vital Signs

Systolic blood pressure, diastolic blood pressure and heart rate etc. and their changes from baseline over time will be summarized by descriptive statistics including mean, standard error etc. Individual subject listing of vital signs will be provided.

## 8.7 Ectopic Mineralization Safety

Ectopic mineralization safety data includes renal ultrasound, ECG, ECHO, serum calcium, creatinine, GFR, iPTH, 24-hr urinary calcium excretion rate, fasting 2-hr urinary calcium/creatinine. The observed values and changes from baseline in the ectopic mineralization safety data will be summarized and listed by individual subjects.

## 8.7.1 Renal Ultrasound

Renal ultrasound will be conducted with findings of nephrocalcinosis graded on a 5-point scale and by a central reader. These results will be summarized by time point. Furthermore, a grade shift table summarizing changes from baseline by time point will also be created.

The number and percentage of subjects with nephrolithiasis observed in the kidney will be summarized by time point. A shift table summarizing changes from baseline by time point will be created.

A listing of renal ultrasound nephrocalcinosis scores, the presence or absence of nephrolithiasis in the kidney and the radiologist's comments will also be provided.

#### 8.7.2 ECG

Descriptive statistics for the absolute measurements and changes from Baseline for selected ECG parameters will be reported. These include the following intervals: QT, QT corrected for heart rate, the time elapsed from the onset of atrial depolarization to the onset of ventricular depolarization (PR), and time elapsed for depolarization of the ventricles (QRS).

The frequency of subjects with a maximum increase from Baseline in the QTc interval will be summarized according to the following categories: >30 ms and >60 ms. In addition, the frequency of subjects with QTc post dose values according to the following categories: >450 ms, >480 ms and >500 ms, will be summarized.

A listing of all ECG parameters including the overall assessment will also be created.

#### 8.7.3 ECHO

ECHO data will be centrally read to assess for evidence of ectopic mineralization in the heart and aorta and to evaluate for signs of LVH or cardiac dysfunction. Descriptive statistics for the various continuous ECHO measurements (e.g., left ventricular mass index, etc.) will be at the scheduled time points and will include the change from baseline value. The summary of



the descriptive statistics will be displayed by visit. Shift tables will be provided for categorical ECHO measurements (e.g. ectopic mineralization score, aortic and mitral valve regurgitation). A listing of all ECHO parameters will be provided.

## 8.8 Endpoints

## 8.8.1 Pharmacodynamic Endpoints

The number and proportion of subjects with serum phosphorus level in the normal range  $(\geq 2.5 \text{ and} < 4.5)$  at each time point will be provided, along with the two-sided 95% confidence intervals, obtained using the GEE model described in Section 8.1.1. An overall summary of the number and proportion of patients who ever reached the normal range over the duration of the study will also be provided. Additional analyses of serum phosphorus including observed values, change from baseline, percent change from baseline over time will be summarized.

For the final analysis, the primary PD endpoints at all post-baseline visits will be compared to baseline using the GEE model described in Section 8.1.1, and the primary statistical comparison will be between the levels at baseline and week 72.

For the interim analysis, the primary PD endpoints at all post-baseline visits prior or at week 24 for all patients will be compared to baseline using the GEE model, and the primary statistical comparison will be between the levels at baseline and week 24.

For all primary PD endpoints descriptive statistics of observed values and of changes from baseline at each visit will be provided.

Graphs showing the change over time in key PD parameter for both observed measure and the change from baseline will be provided. The relationship between various PD parameters as well as KRN23 concentrations may be examined.

#### 8.8.2 Efficacy Endpoints

## 8.8.2.1 PRO Endpoints

BPI (Worst Pain, Pain Severity and Pain Interference), WOMAC (the three domains) and SF-36 (the eight domains and the two components) scores and the proportion of responders at each study time point will be evaluated using descriptive statistics. The binary endpoints (responder/non-responder to treatment) and the changes from baseline to week 24 (interim analysis) and week 72 (final analysis) will be analyzed using the GEE model described in Section 8.1.1. Listings containing the answers to each question and each of the scores over time will also be provided. In addition, the cumulative distribution functions (CDF) based on change from baseline and percent change from baseline of worst Pain score will be provided.



## 8.8.2.2 X-Ray Endpoints

The number, the change from baseline and the location of the active pseudofractures or other disease-related skeletal abnormalities as viewed on standard radiographs at each visit will be evaluated using descriptive statistics. A listing containing the X-Ray endpoints details will also be provided.

#### 8.8.2.3 6-Minute Walk Test and Percent Predicted 6-Minute Walk Test

Summary statistics of total distance walked and percent of predicted 6MWT will be tabulated for each study visit for the observed measures and their respective change from Baseline. Changes from baseline to week 72 will be analyzed using the GEE model described in Section 8.1.1. Changes from baseline to week 24 will be analyzed using paired t-test. A listing containing the 6MWT details will also be provided.

## 8.8.2.4 Timed Up and Go Test

The TUG will be used to evaluate changes in transition time during ambulatory activity that incorporates strength, agility, and dynamic balance. TUG results will be evaluated using descriptive statistics. Changes from baseline to week 72 will be analyzed using the GEE model described in Section 8.1.1. Changes from baseline to week 24 will be analyzed using paired t-test.

A listing containing the TUG details and graphs showing change from baseline in TUG results will be provided.

## 8.8.2.5 Subgroup Analyses

Summary tables for the actual values and change from baseline in:

- BPI scores at each study time point for the subgroups of patients with worst pain score at baseline <4 and ≥4
- SF-36 scores and the proportion of responders at each study time point for the subgroups of patients with baseline PCS T-scores  $\leq 40$  and > 40
- total distance walked and percent of predicted 6MWT for the subgroup of patients with percent predicted 6MWT at baseline  $\leq 80\%$  and > 80%

will be provided.



## 9 REFERENCES

- Bellamy, N. 2012. *WOMAC® Osteoarthritis Index User Guide X*. Brisbane, Australia: University of Queensland.
- Bellamy, N, Wilson, C, and Hendrikz, J. 2011. "Population-based normative values for the Western Ontario and McMaster (WOMAC) Osteoarthritis Index: part I." *Semin Arthritis Rheum* 41 (2):139-48.
- Gibbons, WJ, Fruchter, N, Sloan, S, and Levy, RD. 2001. "Reference values for a multiple repetition 6-minute walk test in healthy adults older than 20 years." *J Cardiopulm.Rehabil.* 21 (2):87-93.
- Maruish, M. 2011. *User's manual for the SF-36v2 Health Survey (3rd ed.)*: Lincoln, RI: QualityMetric Incorporated.

Study Number: UX023-CL203 Statistical Analysis Plan Amendment 1

27 April 2016, Version 1.1



# 10 APPENDICES

# **Appendix 1: UX023-CL203 Efficacy Endpoint Summary Table**

| Test /<br>Instrument | Eligible Study<br>Population | Endpoint | Pharmacodynamics, efficacy<br>or safety endpoint | Timepoints for<br>Assessment | Statistical<br>approach at<br>week 24 analysis | Statistical<br>approach at<br>week 72 analysis |
|---|---|---|---|---|---|---|
| PD | PD PD Analysis Set Change from baseline in serum phosphorus | | Pharmacodynamics | Baseline, Weeks 2, 4, 6, 8, 10, 12, 24, 26, 28, 36, 38, 40 48, 50, 52, 60, 72/ET | GEE Model | GEE Model |
| PD | PD Analysis Set | Percent change from baseline in serum phosphorus | Pharmacodynamics | Baseline, Weeks 2, 4, 6, 8, 10, 12, 24, 26, 28, 36, 38, 40 48, 50, 52, 60, 72/ET | GEE Model | GEE Model |
| PD | PD PD Analysis Set Proportion of subjects with serum phosphorus level in the normal range | | Pharmacodynamics | Baseline, Weeks 2, 4, 6, 8, 10, 12, 24, 26, 28, 36, 38, 40 48, 50, 52, 60, 72/ET | GEE Model | GEE Model |
| PD | PD Analysis Set | Change from baseline in iPTH | Pharmacodynamics | Baseline, Weeks 12, 24, 36, 48, 72 | GEE Model | GEE Model |
| PD | PD Analysis Set | Change from baseline in Total<br>FGF23 | Pharmacodynamics | Baseline, Weeks 4, 8, 12, 24, 28, 36, 40, 48, 72 | GEE Model | GEE Model |
| PD | PD Analysis Set Change from baseline in Free FGF23 | | Pharmacodynamics | Baseline, Weeks 4, 8, 12, 24, 28, 36, 40, 48, 72 | GEE Model | GEE Model |
| PD | PD Analysis Set | Change from baseline in 1,25(OH) <sub>2</sub> D | Pharmacodynamics | Baseline, Weeks 12, 24, 36, 48, 72 | GEE Model | GEE Model |




| Test /<br>Instrument | Eligible Study<br>Population | Endpoint | Pharmacodynamics, efficacy or safety endpoint | Timepoints for<br>Assessment | Statistical<br>approach at<br>week 24 analysis | Statistical<br>approach at<br>week 72 analysis |
|---|---|---|---|---|---|---|
| PD | PD PD Analysis Set Change from baseline in 2 parameters (TmP/GFR, c creatinine, calcium/creatin phosphorus) | | Pharmacodynamics | Baseline, Weeks 12, 24, 36, 48, 72 | GEE Model | GEE Model |
| PD | PD Analysis Set | Change from baseline in 24-hr<br>urine parameters (calcium,<br>calcium/creatinine ratio, creatinine,<br>phosphorus, phosphorus/creatinine<br>ratio) | Pharmacodynamics | Baseline, Weeks 12, 24, 36, 48, 72/ET | GEE Model | GEE Model |
| PD | PD Analysis Set | Change from baseline in fractional excretion of phosphorus | Pharmacodynamics | Baseline, Weeks 12, 24, 36, 48, 72/ET | GEE Model | GEE Model |
| PD | PD Analysis Set | Change from baseline in bone biomarkers (ALP, BALP, CTx, P1NP) | Pharmacodynamics | Baseline, Weeks 24, 48, 72/ET | Paired t-test | GEE Model |
| PD | Safety Analysis<br>Set | Change from baseline in serum calcium | Safety | Baseline, Weeks 2, 4, 6, 8, 10, 12, 24, 26, 28, 36, 38, 40 48, 50, 52, 60, 72/ET | GEE Model | GEE Model |
| PD | Safety Analysis<br>Set | Change from baseline in serum creatinine | Safety | Baseline, Weeks 12, 24, 36, 48, 72/ET | GEE Model | GEE Model |
| PD | Safety Analysis<br>Set | Change from baseline in amylase | Safety | Baseline, Weeks 12, 24, 36, 48, 72/ET | GEE Model | GEE Model |




| Test /<br>Instrument | Eligible Study<br>Population | Endpoint | Pharmacodynamics, efficacy<br>or safety endpoint | Timepoints for<br>Assessment | Statistical<br>approach at<br>week 24 analysis | Statistical<br>approach at<br>week 72 analysis |
|---|---|---|---|---|---|---|
| PD | Safety Analysis<br>Set | Change from baseline in GFR | Safety | Baseline, Weeks 12, 24, 36, 48, 72/ET | GEE Model | GEE Model |
| BPI | Efficacy Analysis<br>Set | Change from baseline in: Worst Pain Pain Severity Pain Interference | Efficacy | Baseline, Weeks 12, 24, 36, 48, 72/ET | GEE Model | GEE Model |
| WOMAC | Efficacy Analysis<br>Set | Change from baseline in: <ul><li>Pain</li><li>Stiffness</li><li>Physical Functioning</li></ul> | Efficacy | Baseline, Weeks 12, 24, 36, 48, 72/ET | GEE Model | GEE Model |
| SF36 | Efficacy Analysis<br>Set | <ul> <li>Change from baseline in:</li> <li>PF, RP, BP, GH, MH, RE, SF,VT scales</li> <li>MCS and PCS summary component scores</li> </ul> | Efficacy | Baseline, Weeks 12, 24, 36, 48, 72/ET | GEE Model | GEE Model |
| 6MWT | Efficacy Analysis<br>Set | Change from baseline in distance traveled during 6 minutes (meters) | Efficacy | Baseline, Weeks 24, 36, 48, 72/ET | Paired t-test | GEE Model |
| 6MWT | Efficacy Analysis<br>Set | Change from baseline in percent predicted of the distance traveled during 6 minutes | Efficacy | Baseline, Weeks 12, 24, 36, 48, 72/ET | Paired t-test | GEE Model |
| TUG | Efficacy Analysis<br>Set | Change from baseline in TUG | Efficacy | Baseline, Weeks 12, 24, 36, 48, 72/ET | Paired t-test | GEE Model |




| Test /<br>Instrument | Eligible Study<br>Population | Endpoint | Pharmacodynamics, efficacy or safety endpoint | Timepoints for<br>Assessment | Statistical<br>approach at<br>week 24 analysis | Statistical<br>approach at<br>week 72 analysis |
|---|---|---|---|---|---|---|
| PD | PD Analysis Set | Change from baseline in chemistry lab parameters (ALT, AST, bilirubin -direct and total, BUN, uric acid, CO <sub>2</sub> , total cholesterol, triglycerides, GGT, glucose, LDH, Potassium, Protein -albumin and total, sodium) | Safety | Baseline, Weeks 12, 24, 36, 48, 72/ET | Descriptive statistics | Descriptive statistics |
| PD | PD Analysis Set | Change from baseline in<br>hematology lab parameters<br>(hematocrit, hemoglobin, platelet,<br>RBC, WBC, MCV, MCH, MCH<br>concentration) | Safety | Baseline, Weeks 12, 24, 36, 48, 72/ET | Descriptive<br>Summary | Descriptive<br>Summary |
| PD | PD Analysis Set | Change from baseline in<br>urinanalysis parameters (pH,<br>ketones, protein, glucose) | Safety | Baseline, Weeks 12, 24, 36, 48, 72/ET | Descriptive<br>Summary | Descriptive<br>Summary |
| ECG | Safety Analysis<br>Set | Change from baseline in ECG parameters (PR, QT, QTc, QRS) | Safety | Baseline, Weeks 24, 48, 72/ET | Descriptive<br>Summary | Descriptive<br>Summary |




# **Appendix 2: BPI Questionnaire**

| | | | Ві | rief F | Pain I | nver | itory | (Sho | rt Fo | orm) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| SUE | BJECT | ID: | | | | | VISIT | DATE | i: | _/ | / |
| 1. | head | aches | | s, and | | | | | | | such as minor<br>an these every- |
| | | | | es/ | | | | | | No | |
| 2. | | ne diag | | nade ir | ı the ar | eas wh | ere you | ı feel p | ain. P | ut an X | on the area that |
| | | | | Right | | eft | Lef | | Right | | |
| 3 | Pleas | se rate | Vour n | ain by | صاب<br>ساب | the or | e numh | oerthat | hest o | escribe | s vour pain at its |
| 3. | worst | in the | last 24 | hours | S. | | | | | | es your pain at its |
| 3. | | | | hours | S. | the or | | | best o | | 10<br>Pain as bad as |
| <ol> <li>3.</li> <li>4.</li> </ol> | 0<br>No<br>Pain | in the | 2 your p | 1 hours 3 ain by | s.<br>4<br>circling | 5 | 6 | 7 | 8 | 9 | 10<br>Pain as bad as |
| | 0<br>No<br>Pain | in the | 2 last 24 | 3 ain by hours | s.<br>4<br>circling | 5 | 6 | 7 | 8 | 9 | 10 Pain as bad as you can imagine as your pain at its 10 Pain as bad as |
| | worst 0 No Pain Pleas least 0 No Pain Pleas | in the 1 se rate in the 1 | e last 24 2 your p last 24 2 your p | 4 hours<br>3<br>ain by<br>hours<br>3 | circling 4 | 5<br>the or<br>5 | 6<br>ne numb<br>6 | 7<br>per that<br>7 | 8<br>best d | 9<br><b>lescribe</b><br>9 | 10 Pain as bad as you can imagine as your pain at its 10 Pain as bad as |
| 4. | worst 0 No Pain Pleas least 0 No Pain Pleas | in the<br>1<br>se rate<br>in the<br>1 | e last 24 2 your p last 24 2 your p | 4 hours<br>3<br>ain by<br>hours<br>3 | circling 4 | 5<br>the or<br>5 | 6<br>ne numb<br>6 | 7<br>per that<br>7 | 8<br>best d | 9<br><b>lescribe</b><br>9 | 10 Pain as bad as you can imagine as your pain at its 10 Pain as bad as you can imagine as your pain on 10 Pain as bad as |
| 4. | worst 0 No Pain Pleast 0 No Pain Pleast the at 0 No Pain | se rate in the 1 se rate verage 1 | e last 24 2 your p last 24 2 your p 2 | ain by hours 3 ain by ain by 3 | circling 4 circling 4 | 5 the or | 6 6 ne numb 6 | 7<br>per that<br>per that<br>7 | 8 8 8 best of | 9<br>lescribe<br>9<br>lescribe | 10 Pain as bad as you can imagine as your pain at its 10 Pain as bad as you can imagine as your pain on |



| SUE | BJECT ID: | | | | | VISIT | DATE: | | ′ | / |
|---|---|---|---|---|---|---|---|---|---|---|
| 7. | What trea | atments o | r med | ications : | are you | receivi | ing for y | our pa | in? | |
| 8. | In the las<br>provided<br>you have | ? Please | circle | | | | | | | |
| | 0% 10%<br>No<br>Relief | 6 20% | 30% | 40% | 50% | 60% | 70% | 80% | 90% | 6 100%<br>Complete<br>Relief |
| 9. | Circle the interfered | | | at descr | ibes ho | w, duri | ng the p | ast 24 | hour | s, pain has |
| | A. Ge | neral Act | ivitv | | | | | | | |
| | 0 1<br>Does not<br>Interfere | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Completely<br>Interferes |
| | B. Mo<br>0 1<br>Does not<br>Interfere | od 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Completely<br>Interferes |
| | C. Wa<br>0 1<br>Does not<br>Interfere | alking Abi<br>2 | lity<br>3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Completely<br>Interferes |
| | D. No | rmal Wor | k (incl | udes bot | h work | outside | the ho | me and | hou | sework) |
| | 0 1<br>Does not<br>Interfere | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Completely<br>Interferes |
| | E. Re | lations wi | th oth | er people | е | | | | | |
| | 0 1<br>Does not<br>Interfere | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Completely<br>Interferes |
| | F. Sle | | | | | | | | | |
| | 0 1<br>Does not<br>Interfere | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Completely<br>Interferes |
| | | oyment c | | | _ | | | | | 40 |
| | 0 1<br>Does not<br>Interfere | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Completely<br>Interferes |
| | | | | | Pain Rese | les S. Clee<br>arch Group<br>reserved | eland, PhD<br>p | | | |
| Pag | e 2 of 2 | | | | | | | | | |



# **Appendix 3: WOMAC Questionnaire**

# WOMAC OSTEOARTHRITIS INDEX VERSION LK3.1 INSTRUCTIONS TO PATIENTS

In Sections A, B, and C questions are asked in the following format. Please select the circle for your response.

| EXAME | PLES: | | | | | |
|---|---|---|---|---|---|---|
| 1. If yo | ou fill in the circ | cle on the fa | r left as shown | below, | | |
| | none | mild | moderate | severe | extreme | |
| ther | n you are indica | ating that yo | u feel <b>no</b> pain. | Ü | | |
| 2. If yo | ou fill in the circ | cle on the fa | r right as showr | n below, | | |
| | none | mild | moderate | severe | extreme<br>• | |
| ther | n you are indica | ating that yo | u feel <b>extreme</b> | pain. | | |
| Please n | ote: | | | | | |
| | | | lect, the <b>more</b> p<br>ect, the <b>less</b> pain | | | |
| | e asked to indica<br>last 48 hours. | ate on this ty | pe of scale the a | mount of pai | n, stiffness or disabili | ty you have felt |
| Which lowe<br>the last 48 | ,, | has been mos | t bothersome and | or has given y | ou the most difficulty i | n |
| | , | | | • | Indicate the severity<br>I feel are caused by the | |



#### Section A PAIN

| Think about the pain you felt in your caused by your arthritis during the <u>last 48 hours</u> . | | | | | |
|---|---|---|---|---|---|
| Question: How much pain have you had | None Mild | | Moderate | Severe | Extreme |
| 1. when walking on a flat surface? | 0 | 0 | 0 | 0 | 0 |
| 2. when going up or down stairs? | 0 | 0 | | | |
| 3. at night while in bed? (that is - pain that disturbs your sleep) | 0 | 0 | 0 | 0 | 0 |
| 4. while sitting or lying down? | 0 | 0 | 0 | 0 | 0 |
| 5. while standing? | 0 | 0 | 0 | 0 | 0 |

## Section B STIFFNESS

| Think about the stiffness (not pain) you felt in your caused by arthritis during the <u>last 48 hours</u> . Stiffness is a sensation of <b>decreased</b> ease in moving your joint. | | | | | |
|---|---|---|---|---|---|
| | None | Mild | Moderate | Severe | Extreme |
| 6. How <b>severe</b> has your stiffness been <b>after you first woke up</b> in the morning? | 0 | 0 | 0 | | 0 |
| 7. How <b>severe</b> has your stiffness been after sitting or lying down or while resting <b>later in the day</b> ? | 0 | | 0 | 0 | 0 |


## Section C DIFFICULTY PERFORMING DAILY ACTIVITIES

| Think about the difficulty you had in doing the following daily physical activities caused by the arthritis in yourduring the <u>last 48 hours</u> . By this we mean <b>your ability to move around and take care of yourself.</b> | | | | | |
|---|---|---|---|---|---|
| Question: How much difficulty have you had | None | Mild | Moderate | Severe | Extreme |
| 8. when going down the stairs? | 0 | 0 | 0 | 0 | 0 |
| 9. when going up the stairs? | | | 0 | 0 | 0 |
| 10. when getting up from a sitting position? | 0 | 0 | 0 | 0 | 0 |
| 11. while standing? | | 0 | 0 | 0 | 0 |
| 12. when bending to the floor? | | 0 | 0 | | 0 |
| 13. when walking on a flat surface? | | | 0 | | 0 |
| 14. getting in or out of a car, or getting on or off a bus? | | 0 | | | |
| 15. while going shopping? | 0 | | 0 | | 0 |
| 16. when putting on your socks or panty hose or stockings? | | 0 | 0 | 0 | 0 |
| 17. when getting out of bed? | | 0 | 0 | 0 | 0 |
| 18. when taking off your socks or panty hose or stockings? | | 0 | 0 | 0 | 0 |
| 19. while lying in bed? | 0 | 0 | 0 | 0 | 0 |
| 20. when getting in or out of the bathtub? | | | 0 | | |
| 21. while sitting? | | 0 | 0 | | |
| 22. when getting on or off the toilet? | | | 0 | | 0 |
| 23. while doing heavy household chores? | 0 | 0 | 0 | 0 | 0 |
| 24. while doing light household chores? | | 0 | 0 | 0 | 0 |



#### **Appendix 4: SF-36 Questionnaire**

# Your Health and Well-Being

This survey asks for your views about your health. This information will help keep track of how you feel and how well you are able to do your usual activities. Thank you for completing this survey!

For each of the following questions, please mark an  $\boxtimes$  in the one box that best describes your answer.

1. In general, would you say your health is:

| | Excellent | Very good | Good | Fair | Poor |
|---|------------|------------|------------|------------|------------|
| ' | lacksquare | lacksquare | lacksquare | lacksquare | lacksquare |
| | 1 | 2 | 3 | 4 | 5 |

2. Compared to one year ago, how would you rate your health in general now?

| Much better<br>now than one<br>year ago | Somewhat<br>better<br>now than one<br>year ago | About the same as one year ago | Somewhat<br>worse<br>now than one<br>year ago | Much worse<br>now than one<br>year ago |
|---|---|---|---|---|
| lacktriangle | lacksquare | lacktriangle | lacksquare | lacksquare |
| 1 | 2 | 3 | 4 | 5 |



3. The following questions are about activities you might do during a typical day. Does your health now limit you in these activities? If so, how much?

| | | Yes,<br>limited<br>a lot | Yes,<br>limited<br>a little | No, not<br>limited<br>at all |
|---|---|---|---|---|
| 2 | Vigorous activities, such as running, lifting heavy objects, participating in strenuous sports | 1 | 2 | 3 |
| ь | Moderate activities, such as moving a table, pushing a vacuum cleaner, bowling, or playing golf | 1 | 2 | 3 |
| c | Lifting or carrying groceries | 1 | 2 | 3 |
| d | Climbing several flights of stairs | 1 | 2 | 3 |
| ۰ | Climbing one flight of stairs | 1 | 2 | 3 |
| f | Bending, kneeling, or stooping | 1 | 2 | 3 |
| g | Walking more than a mile | 1 | 2 | 3 |
| h | Walking several hundred yards | 1 | 2 | 3 |
| i | Walking one hundred yards | 1 | 2 | 3 |
| j | Bathing or dressing yourself | 1 | 2 | 3 |



4. During the <u>past 4 weeks</u>, how much of the time have you had any of the following problems with your work or other regular daily activities <u>as a result of your physical health?</u>

| | | All of<br>the time | Most of<br>the time | Some of<br>the time | A little of<br>the time | None of<br>the time |
|---|---|---|---|---|---|---|
| 3 | Cut down on the <u>amount of</u><br>time you spent on work or<br>other activities | <b>▼</b> | <b>▼</b> | | □ 4 | <b>▼</b> |
| ъ | Accomplished less than you would like | 1 | 2 | 3 | 4 | 5 |
| c | Were limited in the <u>kind</u> of work or other activities | 1 | 2 | 3 | 4 | 5 |
| d | Had <u>difficulty</u> performing the work or other activities (for example, it took extra effort) | 1 | 2 | 3 | 4 | 5 |
| 5. | During the past 4 weeks, | how much | of the time | havo von | | |
| | following problems with result of any emotional p | your work | or other re | gular daily | activities : | as a |
| | | your work | or other re ich as feeli Most of | gular daily<br>ng depress | activities : | as a |
| a | | your work roblems (su All of the time | or other re ich as feeli Most of | gular daily<br>ng depress<br>Some of | A little of the time | us)? None of |
| | Cut down on the amount of time you spent on work or | your work roblems (su All of the time | or other re ich as feeli Most of | Some of the time | A little of the time | us)? None of |

SF-36v2\* Health Survey © 1992, 1996, 2000 Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved. SF-36\* is a registered trademark of Medical Outcomes Trust. (SF-36v2\* Health Survey Standard, United States (English))



6. During the <u>past 4 weeks</u>, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups?



7. How much bodily pain have you had during the past 4 weeks?

| None | Very mild | Mild | Moderate | Severe | Very severe |
|------|-----------|------|----------|--------|-------------|
| _ 1 | 2 | 3 | 4 | 5 | 6 |

8. During the <u>past 4 weeks</u>, how much did <u>pain</u> interfere with your normal work (including both work outside the home and housework)?

| Not at all | A little bit | Moderately | Quite a bit | Extremely |
|------------|--------------|------------|-------------|-----------|
| _ 1 | 2 | 3 | 4 | 5 |



9. These questions are about how you feel and how things have been with you during the past 4 weeks. For each question, please give the one answer that comes closest to the way you have been feeling. How much of the time during the past 4 weeks...

| | | All of<br>the time | Most of<br>the time | Some of<br>the time | A little of the time | None of<br>the time |
|---|---|---|---|---|---|---|
| | | | | | • | |
| a | Did you feel full of life? | 1 | 2 | 3 | 4 | 5 |
| ь | Have you been very nervous? | 1 | 2 | 3 | 4 | 5 |
| c | Have you felt so down in the dumps that nothing could cheer you up? | 1 | 2 | 3 | 4 | 5 |
| d | Have you felt calm and peaceful? | 1 | 2 | 3 | 4 | 5 |
| ۰ | Did you have a lot of energy? | 1 | 2 | 3 | 4 | 5 |
| f | Have you felt downhearted and depressed? | 1 | 2 | 3 | 4 | 5 |
| 8 | Did you feel worn out? | 1 | 2 | 3 | 4 | 5 |
| h | Have you been happy? | 1 | 2 | 3 | 4 | 5 |
| i | Did you feel tired? | 1 | 2 | 3 | 4 | 5 |
| 10. | During the past 4 weeks, lemotional problems interfriends, relatives, etc.)? All of Most of the time the time | fered with | your social | • | (like visiting | |
| | the time the time | e the | time t | ine time | the time | |
| | | Γ | ] 3 | □ 4 | □ 5 | |

SF-36v2® Health Survey © 1992, 1996, 2000 Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved. SF-36® is a registered trademark of Medical Outcomes Trust. (SF-36v2® Health Survey Standard, United States (English))



#### 11. How TRUE or FALSE is each of the following statements for you?

| | | Definitely true | Mostly<br>true | Don't<br>know | Mostly false | Definitely false |
|---|---|---|---|---|---|---|
| a | I seem to get sick a little<br>easier than other people | 🗌 1 | 2 | ] з | 4 | 5 |
| ь | I am as healthy as<br>anybody I know | 🗌 1 | 2 | 3 | 4 | 5 |
| с | I expect my health to get worse | 1 | 2 | 3 | 4 | 5 |
| d | My health is excellent | 1 | 2 | 3 | | 5 |

Thank you for completing these questions!



#### **Appendix 5: Events to Monitor**

Injection site reactions: based on HLT "Injection site reaction"

| Category | PT |
|-------------------------|----------------------------------|
| Injection site reaction | Embolia cutis medicamentosa |
| Injection site reaction | Injected limb mobility decreased |
| Injection site reaction | Injection site abscess |
| Injection site reaction | Injection site abscess sterile |
| Injection site reaction | Injection site anaesthesia |
| Injection site reaction | Injection site atrophy |
| Injection site reaction | Injection site bruising |
| Injection site reaction | Injection site calcification |
| Injection site reaction | Injection site cellulitis |
| Injection site reaction | Injection site coldness |
| Injection site reaction | Injection site cyst |
| Injection site reaction | Injection site dermatitis |
| Injection site reaction | Injection site discharge |
| Injection site reaction | Injection site discolouration |
| Injection site reaction | Injection site discomfort |
| Injection site reaction | Injection site dryness |
| Injection site reaction | Injection site dysaesthesia |
| Injection site reaction | Injection site eczema |
| Injection site reaction | Injection site erosion |
| Injection site reaction | Injection site erythema |
| Injection site reaction | Injection site exfoliation |
| Injection site reaction | Injection site extravasation |
| Injection site reaction | Injection site fibrosis |
| Injection site reaction | Injection site granuloma |
| Injection site reaction | Injection site haematoma |
| Injection site reaction | Injection site haemorrhage |
| Injection site reaction | Injection site hyperaesthesia |
| Injection site reaction | Injection site hypersensitivity |
| Injection site reaction | Injection site hypertrichosis |
| Injection site reaction | Injection site hypertrophy |
| Injection site reaction | Injection site hypoaesthesia |
| Injection site reaction | Injection site induration |
| Injection site reaction | Injection site infection |
| Injection site reaction | Injection site inflammation |
| Injection site reaction | Injection site injury |
| Injection site reaction | Injection site irritation |
| Injection site reaction | Injection site ischaemia |
| Injection site reaction | Injection site joint discomfort |



| Category | PT |
|-------------------------|------------------------------------------|
| Injection site reaction | Injection site joint effusion |
| Injection site reaction | Injection site joint erythema |
| Injection site reaction | Injection site joint infection |
| Injection site reaction | Injection site joint inflammation |
| Injection site reaction | Injection site joint movement impairment |
| Injection site reaction | Injection site joint pain |
| Injection site reaction | Injection site joint swelling |
| Injection site reaction | Injection site joint warmth |
| Injection site reaction | Injection site laceration |
| Injection site reaction | Injection site lymphadenopathy |
| Injection site reaction | Injection site macule |
| Injection site reaction | Injection site mass |
| Injection site reaction | Injection site movement impairment |
| Injection site reaction | Injection site necrosis |
| Injection site reaction | Injection site nerve damage |
| Injection site reaction | Injection site nodule |
| Injection site reaction | Injection site oedema |
| Injection site reaction | Injection site pain |
| Injection site reaction | Injection site pallor |
| Injection site reaction | Injection site papule |
| Injection site reaction | Injection site paraesthesia |
| Injection site reaction | Injection site phlebitis |
| Injection site reaction | Injection site photosensitivity reaction |
| Injection site reaction | Injection site plaque |
| Injection site reaction | Injection site pruritus |
| Injection site reaction | Injection site pustule |
| Injection site reaction | Injection site rash |
| Injection site reaction | Injection site reaction |
| Injection site reaction | Injection site recall reaction |
| Injection site reaction | Injection site scab |
| Injection site reaction | Injection site scar |
| Injection site reaction | Injection site streaking |
| Injection site reaction | Injection site swelling |
| Injection site reaction | Injection site thrombosis |
| Injection site reaction | Injection site ulcer |
| Injection site reaction | Injection site urticaria |
| Injection site reaction | Injection site vasculitis |
| Injection site reaction | Injection site vesicles |
| Injection site reaction | Injection site warmth |
| Injection site reaction | Malabsorption from injection site |



Immunogenicity: based on relevant PTs in the narrow SMQs for "Hypersensitivity",

| Category | PT |
|------------------|--------------------------------------------|
| Hypersensitivity | Acute generalised exanthematous pustulosis |
| Hypersensitivity | Administration site dermatitis |
| Hypersensitivity | Administration site eczema |
| Hypersensitivity | Administration site hypersensitivity |
| Hypersensitivity | Administration site rash |
| Hypersensitivity | Administration site recall reaction |
| Hypersensitivity | Administration site urticaria |
| Hypersensitivity | Administration site vasculitis |
| Hypersensitivity | Allergic bronchitis |
| Hypersensitivity | Allergic colitis |
| Hypersensitivity | Allergic cough |
| Hypersensitivity | Allergic cystitis |
| Hypersensitivity | Allergic eosinophilia |
| Hypersensitivity | Allergic gastroenteritis |
| Hypersensitivity | Allergic granulomatous angiitis |
| Hypersensitivity | Allergic hepatitis |
| Hypersensitivity | Allergic keratitis |
| Hypersensitivity | Allergic myocarditis |
| Hypersensitivity | Allergic oedema |
| Hypersensitivity | Allergic otitis externa |
| Hypersensitivity | Allergic otitis media |
| Hypersensitivity | Allergic pharyngitis |
| Hypersensitivity | Allergic respiratory disease |
| Hypersensitivity | Allergic respiratory symptom |
| Hypersensitivity | Allergic sinusitis |
| Hypersensitivity | Allergic transfusion reaction |
| Hypersensitivity | Allergy alert test positive |
| Hypersensitivity | Allergy test positive |
| Hypersensitivity | Allergy to immunoglobulin therapy |
| Hypersensitivity | Allergy to vaccine |
| Hypersensitivity | Alveolitis allergic |
| Hypersensitivity | Anaphylactic reaction |
| Hypersensitivity | Anaphylactic shock |
| Hypersensitivity | Anaphylactic transfusion reaction |
| Hypersensitivity | Anaphylactoid reaction |
| Hypersensitivity | Anaphylactoid shock |
| Hypersensitivity | Anaphylaxis treatment |
| Hypersensitivity | Angioedema |



| Category | PT |
|------------------|----------------------------------------------------------|
| Hypersensitivity | Antiallergic therapy |
| Hypersensitivity | Antiendomysial antibody positive |
| Hypersensitivity | Anti-neutrophil cytoplasmic antibody positive vasculitis |
| Hypersensitivity | Application site dermatitis |
| Hypersensitivity | Application site eczema |
| Hypersensitivity | Application site hypersensitivity |
| Hypersensitivity | Application site rash |
| Hypersensitivity | Application site recall reaction |
| Hypersensitivity | Application site urticaria |
| Hypersensitivity | Application site vasculitis |
| Hypersensitivity | Arthritis allergic |
| Hypersensitivity | Atopy |
| Hypersensitivity | Blepharitis allergic |
| Hypersensitivity | Blood immunoglobulin E abnormal |
| Hypersensitivity | Blood immunoglobulin E increased |
| Hypersensitivity | Bromoderma |
| Hypersensitivity | Bronchospasm |
| Hypersensitivity | Catheter site dermatitis |
| Hypersensitivity | Catheter site eczema |
| Hypersensitivity | Catheter site hypersensitivity |
| Hypersensitivity | Catheter site rash |
| Hypersensitivity | Catheter site urticaria |
| Hypersensitivity | Catheter site vasculitis |
| Hypersensitivity | Chronic eosinophilic rhinosinusitis |
| Hypersensitivity | Chronic hyperplastic eosinophilic sinusitis |
| Hypersensitivity | Circulatory collapse |
| Hypersensitivity | Circumoral oedema |
| Hypersensitivity | Conjunctival oedema |
| Hypersensitivity | Conjunctivitis allergic |
| Hypersensitivity | Corneal oedema |
| Hypersensitivity | Cutaneous vasculitis |
| Hypersensitivity | Dennie-Morgan fold |
| Hypersensitivity | Dermatitis |
| Hypersensitivity | Dermatitis acneiform |
| Hypersensitivity | Dermatitis allergic |
| Hypersensitivity | Dermatitis atopic |
| Hypersensitivity | Dermatitis bullous |
| Hypersensitivity | Dermatitis contact |
| Hypersensitivity | Dermatitis exfoliative |
| Hypersensitivity | Dermatitis exfoliative generalised |



| Category | PT |
|------------------|-------------------------------------------------------|
| Hypersensitivity | Dermatitis herpetiformis |
| Hypersensitivity | Dermatitis infected |
| Hypersensitivity | Dermatitis psoriasiform |
| Hypersensitivity | Distributive shock |
| Hypersensitivity | Documented hypersensitivity to administered product |
| Hypersensitivity | Drug cross-reactivity |
| Hypersensitivity | Drug eruption |
| Hypersensitivity | Drug hypersensitivity |
| Hypersensitivity | Drug provocation test |
| Hypersensitivity | Drug reaction with eosinophilia and systemic symptoms |
| Hypersensitivity | Eczema |
| Hypersensitivity | Eczema infantile |
| Hypersensitivity | Eczema nummular |
| Hypersensitivity | Eczema vaccinatum |
| Hypersensitivity | Eczema vesicular |
| Hypersensitivity | Eczema weeping |
| Hypersensitivity | Encephalitis allergic |
| Hypersensitivity | Encephalopathy allergic |
| Hypersensitivity | Epidermal necrosis |
| Hypersensitivity | Epidermolysis |
| Hypersensitivity | Epidermolysis bullosa |
| Hypersensitivity | Epiglottic oedema |
| Hypersensitivity | Erythema multiforme |
| Hypersensitivity | Erythema nodosum |
| Hypersensitivity | Exfoliative rash |
| Hypersensitivity | Eye allergy |
| Hypersensitivity | Eye oedema |
| Hypersensitivity | Eye swelling |
| Hypersensitivity | Eyelid oedema |
| Hypersensitivity | Face oedema |
| Hypersensitivity | Giant papillary conjunctivitis |
| Hypersensitivity | Gingival oedema |
| Hypersensitivity | Gingival swelling |
| Hypersensitivity | Gleich's syndrome |
| Hypersensitivity | Haemorrhagic urticaria |
| Hypersensitivity | Hand dermatitis |
| Hypersensitivity | Henoch-Schonlein purpura |
| Hypersensitivity | Henoch-Schonlein purpura nephritis |
| Hypersensitivity | Hereditary angioedema |
| Hypersensitivity | Hypersensitivity |



| Category | PT |
|------------------|---------------------------------------|
| Hypersensitivity | Hypersensitivity vasculitis |
| Hypersensitivity | Idiopathic urticaria |
| Hypersensitivity | Immediate post-injection reaction |
| Hypersensitivity | Immune thrombocytopenic purpura |
| Hypersensitivity | Immune tolerance induction |
| Hypersensitivity | Infusion site dermatitis |
| Hypersensitivity | Infusion site eczema |
| Hypersensitivity | Infusion site hypersensitivity |
| Hypersensitivity | Infusion site rash |
| Hypersensitivity | Infusion site recall reaction |
| Hypersensitivity | Infusion site urticaria |
| Hypersensitivity | Infusion site vasculitis |
| Hypersensitivity | Injection site dermatitis |
| Hypersensitivity | Injection site eczema |
| Hypersensitivity | Injection site hypersensitivity |
| Hypersensitivity | Injection site rash |
| Hypersensitivity | Injection site recall reaction |
| Hypersensitivity | Injection site urticaria |
| Hypersensitivity | Injection site vasculitis |
| Hypersensitivity | Instillation site hypersensitivity |
| Hypersensitivity | Instillation site rash |
| Hypersensitivity | Instillation site urticaria |
| Hypersensitivity | Interstitial granulomatous dermatitis |
| Hypersensitivity | Intestinal angioedema |
| Hypersensitivity | Iodine allergy |
| Hypersensitivity | Kaposi's varicelliform eruption |
| Hypersensitivity | Kounis syndrome |
| Hypersensitivity | Laryngeal oedema |
| Hypersensitivity | Laryngitis allergic |
| Hypersensitivity | Laryngospasm |
| Hypersensitivity | Laryngotracheal oedema |
| Hypersensitivity | Limbal swelling |
| Hypersensitivity | Lip oedema |
| Hypersensitivity | Lip swelling |
| Hypersensitivity | Mast cell degranulation present |
| Hypersensitivity | Mouth swelling |
| Hypersensitivity | Mucocutaneous rash |
| Hypersensitivity | Multiple allergies |
| Hypersensitivity | Nephritis allergic |
| Hypersensitivity | Nikolsky's sign |



| Category | PT |
|------------------|-------------------------------------------------|
| Hypersensitivity | Nodular rash |
| Hypersensitivity | Oculomucocutaneous syndrome |
| Hypersensitivity | Oculorespiratory syndrome |
| Hypersensitivity | Oedema mouth |
| Hypersensitivity | Oral allergy syndrome |
| Hypersensitivity | Oropharyngeal blistering |
| Hypersensitivity | Oropharyngeal spasm |
| Hypersensitivity | Oropharyngeal swelling |
| Hypersensitivity | Palatal oedema |
| Hypersensitivity | Palatal swelling |
| Hypersensitivity | Palisaded neutrophilic granulomatous dermatitis |
| Hypersensitivity | Palpable purpura |
| Hypersensitivity | Pathergy reaction |
| Hypersensitivity | Periorbital oedema |
| Hypersensitivity | Pharyngeal oedema |
| Hypersensitivity | Pruritus allergic |
| Hypersensitivity | Radioallergosorbent test positive |
| Hypersensitivity | Rash |
| Hypersensitivity | Rash erythematous |
| Hypersensitivity | Rash follicular |
| Hypersensitivity | Rash generalised |
| Hypersensitivity | Rash macular |
| Hypersensitivity | Rash maculo-papular |
| Hypersensitivity | Rash maculovesicular |
| Hypersensitivity | Rash morbilliform |
| Hypersensitivity | Rash neonatal |
| Hypersensitivity | Rash papulosquamous |
| Hypersensitivity | Rash pruritic |
| Hypersensitivity | Rash pustular |
| Hypersensitivity | Rash rubelliform |
| Hypersensitivity | Rash scarlatiniform |
| Hypersensitivity | Rash vesicular |
| Hypersensitivity | Reaction to azo-dyes |
| Hypersensitivity | Reaction to colouring |
| Hypersensitivity | Reaction to drug excipients |
| Hypersensitivity | Reaction to preservatives |
| Hypersensitivity | Red man syndrome |
| Hypersensitivity | Rhinitis allergic |
| Hypersensitivity | Scleral oedema |
| Hypersensitivity | Scleritis allergic |



| Category | PT |
|------------------|-------------------------------------------|
| Hypersensitivity | Scrotal oedema |
| Hypersensitivity | Serum sickness |
| Hypersensitivity | Serum sickness-like reaction |
| Hypersensitivity | Shock |
| Hypersensitivity | Shock symptom |
| Hypersensitivity | Skin necrosis |
| Hypersensitivity | Skin reaction |
| Hypersensitivity | Skin test positive |
| Hypersensitivity | Solar urticaria |
| Hypersensitivity | Solvent sensitivity |
| Hypersensitivity | Stevens-Johnson syndrome |
| Hypersensitivity | Stoma site hypersensitivity |
| Hypersensitivity | Stoma site rash |
| Hypersensitivity | Swelling face |
| Hypersensitivity | Swollen tongue |
| Hypersensitivity | Tongue oedema |
| Hypersensitivity | Toxic epidermal necrolysis |
| Hypersensitivity | Toxic skin eruption |
| Hypersensitivity | Tracheal oedema |
| Hypersensitivity | Type I hypersensitivity |
| Hypersensitivity | Type II hypersensitivity |
| Hypersensitivity | Type III immune complex mediated reaction |
| Hypersensitivity | Type IV hypersensitivity reaction |
| Hypersensitivity | Urticaria |
| Hypersensitivity | Urticaria cholinergic |
| Hypersensitivity | Urticaria chronic |
| Hypersensitivity | Urticaria contact |
| Hypersensitivity | Urticaria papular |
| Hypersensitivity | Urticaria physical |
| Hypersensitivity | Urticaria pigmentosa |
| Hypersensitivity | Urticaria vesiculosa |
| Hypersensitivity | Vaginal exfoliation |
| Hypersensitivity | Vaginal ulceration |
| Hypersensitivity | Vasculitic rash |
| Hypersensitivity | Vessel puncture site rash |
| Hypersensitivity | Vulval ulceration |
| Hypersensitivity | Vulvovaginal rash |
| Hypersensitivity | Vulvovaginal ulceration |



Hyperphosphataemia: based on selected PTs below

| Category | PT |
|--------------------|----------------------------|
| Hyperphosphataemia | Hyperphosphataemia |
| Hyperphosphataemia | Blood phosphorus increased |

Ectopic mineralization: based on a MedDRA search of 'calcification'

| Category | PT |
|-----------------------|-----------------------------------|
| Ectopic calcification | Adrenal calcification |
| Ectopic calcification | Aortic calcification |
| Ectopic calcification | Aortic valve calcification |
| Ectopic calcification | Aortic valve sclerosis |
| Ectopic calcification | Articular calcification |
| Ectopic calcification | Bladder wall calcification |
| Ectopic calcification | Breast calcifications |
| Ectopic calcification | Bursa calcification |
| Ectopic calcification | Calcific deposits removal |
| Ectopic calcification | Calcification metastatic |
| Ectopic calcification | Calcification of muscle |
| Ectopic calcification | Calcinosis |
| Ectopic calcification | Calculus bladder |
| Ectopic calcification | Calculus prostatic |
| Ectopic calcification | Calculus ureteric |
| Ectopic calcification | Calculus urethral |
| Ectopic calcification | Calculus urinary |
| Ectopic calcification | Cardiac valve sclerosis |
| Ectopic calcification | Cerebral calcification |
| Ectopic calcification | Chondrocalcinosis |
| Ectopic calcification | Chondrocalcinosis pyrophosphate |
| Ectopic calcification | Cutaneous calcification |
| Ectopic calcification | Dystrophic calcification |
| Ectopic calcification | Heart valve calcification |
| Ectopic calcification | Heart valve stenosis |
| Ectopic calcification | Hepatic calcification |
| Ectopic calcification | Intervertebral disc calcification |
| Ectopic calcification | Intestinal calcification |
| Ectopic calcification | Ligament calcification |
| Ectopic calcification | Lymph node calcification |
| Ectopic calcification | Mitral valve calcification |
| Ectopic calcification | Mitral valve sclerosis |
| Ectopic calcification | Myocardial calcification |



| Category | PT |
|---|---|
| Ectopic calcification | Nephrocalcinosis |
| Ectopic calcification | Nephrolithiasis |
| Ectopic calcification | Ovarian calcification |
| Ectopic calcification | Pancreatic calcification |
| Ectopic calcification | Pericardial calcification |
| Ectopic calcification | Pleural calcification |
| Ectopic calcification | Prostatic calcification |
| Ectopic calcification | Pulmonary calcification |
| Ectopic calcification | Pulmonary valve calcification |
| Ectopic calcification | Pulmonary valve sclerosis |
| Ectopic calcification | Splenic calcification |
| Ectopic calcification | Stag horn calculus |
| Ectopic calcification | Tendon calcification |
| Ectopic calcification | Tracheal calcification |
| Ectopic calcification | Tricuspid valve calcification |
| Ectopic calcification | Tricuspid valve sclerosis |
| Ectopic calcification | Vascular calcification |

Gastrointestinal: based on narrow SMQ "Gastrointestinal nonspecific inflammation and dysfunctional conditions"

| Category | PT |
|---|---|
| Gastrointestinal | Acid peptic disease |
| Gastrointestinal | Duodenogastric reflux |
| Gastrointestinal | Dyspepsia |
| Gastrointestinal | Gastrooesophageal reflux disease |
| Gastrointestinal | Gastrooesophageal sphincter insufficiency |
| Gastrointestinal | Chronic gastritis |
| Gastrointestinal | Colitis |
| Gastrointestinal | Duodenitis |
| Gastrointestinal | Enteritis |
| Gastrointestinal | Erosive duodenitis |
| Gastrointestinal | Erosive oesophagitis |
| Gastrointestinal | Feline oesophagus |
| Gastrointestinal | Functional gastrointestinal disorder |
| Gastrointestinal | Gastric mucosa erythema |
| Gastrointestinal | Gastritis |
| Gastrointestinal | Gastritis erosive |
| Gastrointestinal | Gastroduodenitis |
| Gastrointestinal | Gastrointestinal erosion |
| Gastrointestinal | Gastrointestinal mucosa hyperaemia |



| Category | PT |
|------------------|--------------------------------------|
| Gastrointestinal | Gastrointestinal mucosal exfoliation |
| Gastrointestinal | Haemorrhagic erosive gastritis |
| Gastrointestinal | Intestinal angioedema |
| Gastrointestinal | Oesophageal mucosa erythema |
| Gastrointestinal | Oesophagitis |
| Gastrointestinal | Reactive gastropathy |
| Gastrointestinal | Reflux gastritis |
| Gastrointestinal | Remnant gastritis |
| Gastrointestinal | Ulcerative gastritis |
| Gastrointestinal | Abdominal discomfort |
| Gastrointestinal | Abdominal distension |
| Gastrointestinal | Abdominal pain |
| Gastrointestinal | Abdominal pain lower |
| Gastrointestinal | Abdominal pain upper |
| Gastrointestinal | Abdominal symptom |
| Gastrointestinal | Abdominal tenderness |
| Gastrointestinal | Abnormal faeces |
| Gastrointestinal | Aerophagia |
| Gastrointestinal | Anorectal discomfort |
| Gastrointestinal | Bowel movement irregularity |
| Gastrointestinal | Change of bowel habit |
| Gastrointestinal | Constipation |
| Gastrointestinal | Defaecation urgency |
| Gastrointestinal | Diarrhoea |
| Gastrointestinal | Epigastric discomfort |
| Gastrointestinal | Eructation |
| Gastrointestinal | Faecal volume decreased |
| Gastrointestinal | Faecal volume increased |
| Gastrointestinal | Faeces hard |
| Gastrointestinal | Faeces soft |
| Gastrointestinal | Flatulence |
| Gastrointestinal | Frequent bowel movements |
| Gastrointestinal | Gastrointestinal pain |
| Gastrointestinal | Gastrointestinal sounds abnormal |
| Gastrointestinal | Gastrointestinal toxicity |
| Gastrointestinal | Infrequent bowel movements |
| Gastrointestinal | Nausea |
| Gastrointestinal | Non-cardiac chest pain |
| Gastrointestinal | Oesophageal discomfort |
| Gastrointestinal | Oesophageal pain |
| Gastrointestinal | Vomiting |



#### Restless legs syndrome:

| Category | PT |
|------------------------|---------------------------|
| Restless legs syndrome | Restless legs syndrome |
| Restless legs syndrome | Restlessness |
| Restless legs syndrome | Akathisia |
| Restless legs syndrome | Psychomotor hyperactivity |
| Restless legs syndrome | Sensory disturbance |
| Restless legs syndrome | Muscle cramp |
| Restless legs syndrome | Limb discomfort |
| Restless legs syndrome | Neuromuscular pain |
| Restless legs syndrome | Formication |



### **Appendix 6: Schedule of Events**

| VISIT TYPE / NUMBER | Scr <sup>1</sup> | BL <sup>2</sup> 2 | НН <sup>3</sup><br>3 | 4 | НН <sup>3</sup><br>5 | 6 | НН <sup>3</sup><br>7 | 8 | НН <sup>3</sup><br>9 | HH <sup>3</sup><br>10 | 11 | HH <sup>3</sup> | НН <sup>3</sup><br>13 | НН <sup>3</sup><br>14 | 15 | НН <sup>3</sup><br>16 | HH <sup>3</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| WEEK <sup>4</sup> | D-1 | 0 | 2 | 4 | 6 | 8 | 10 | 12 | 16 | 20 | 24 | 26 | 28 | 32 | 36 | 38 | 40 |
| Informed Consent | X | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion<br>Criteria | X | | | | | | | | | | | | | | | | |
| Medical History & Demographics <sup>5</sup> | X | | | | | | | | | | | | | | | | |
| Renal Ultrasound | X | | | | | | | | | | X | | | | | | |
| Chemistry <sup>6</sup> , Hematology <sup>7</sup> ,<br>Urinalysis | X | | | | | | | X | | | X | | | | X | | |
| 2-hr and 24-hr Urine | X | | | | | | | X | | | X | | | | X | | |
| Urine Pregnancy Test <sup>8</sup> | X | X | | X | | X | | X | X | X | X | | X | X | X | | X |
| Vital Signs <sup>9</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Height | | X | | | | | | | | | X | | | | X | | |
| Physical Examination | | X | | | | | | X | | | X | | | | X | | |
| PHEX mutation analysis | | X | | | | | | | | | | | | | | | |
| Anti-KRN23 antibody (HAHA) <sup>10</sup> | | X | | X | | | | X | | | X | | | | X | | |
| Serum Phosphorus | X | X | X | X <sup>11</sup> | X | X <sup>11</sup> | X | X <sup>11</sup> | | | X | X | X | | X | X | X |
| Serum Calcium | X | X | X | X | X | X | X | X | | | X | X | X | | X | X | X |
| Serum Creatinine | X | | | | | | | X | | | X | | | | X | | |
| Serum iPTH | | X | | | | | | X | | | X | | | | X | | |
| Serum FGF23 | | X | | X | | X | | X | | | X | | X | | X | | X |




| VISIT TYPE / NUMBER | Scr <sup>1</sup> | BL <sup>2</sup><br>2 | НН <sup>3</sup> | 4 | НН <sup>3</sup><br>5 | 6 | НН <sup>3</sup><br>7 | 8 | НН <sup>3</sup><br>9 | НН <sup>3</sup><br>10 | 11 | НН <sup>3</sup><br>12 | НН <sup>3</sup><br>13 | НН <sup>3</sup><br>14 | 15 | НН <sup>3</sup><br>16 | НН <sup>3</sup><br>17 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| WEEK <sup>4</sup> | D-1 | 0 | 2 | 4 | 6 | 8 | 10 | 12 | 16 | 20 | 24 | 26 | 28 | 32 | 36 | 38 | 40 |
| Serum 1,25(OH) <sub>2</sub> D | | X | | | | | | X | | | X | | | | X | | |
| Bone Biomarkers <sup>12</sup> | | X | | | | | | | | | X | | | | | | |
| ECHO, ECG | | X | | | | | | | | | X | | | | | | |
| WOMAC, BPI, SF36 <sup>13</sup> | | X | | | | | | X | | | X | | | | X | | |
| 6MWT, 3MSCT, TUG | | X | | | | | | | | | X | | | | X | | |
| X-Ray <sup>14</sup> | | X | | | | | | X | | | X | | | | X | | |
| Interval History | | | | | | | | X | | | X | | | | X | | |
| Prior and Concomitant<br>Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Weight | | X | | X | | X | | X | | | X | | | | X | | |
| Drug Administration | | X | | X | | X | | X | X | X | X | | X | X | X | | X |




| VISIT TYPE / NUMBER | HH <sup>3</sup> 18 | 19 | HH <sup>3</sup> 20 | HH <sup>3</sup><br>21 | HH <sup>3</sup> 22 | HH <sup>3</sup> 23 | HH <sup>3</sup> 24 | HH <sup>3</sup> 25 | 26 |
|---|---|---|---|---|---|---|---|---|---|
| WEEK <sup>4</sup> | 44 | 48 | 50 | 52 | 56 | 60 | 64 | 68 | 72/<br>EoT <sup>15</sup> |
| Informed Consent | | | | | | | | | |
| Inclusion/Exclusion Criteria | | | | | | | | | |
| Medical History & Demographics <sup>5</sup> | | | | | | | | | |
| Renal Ultrasound | | X | | | | | | | X |
| Chemistry <sup>6</sup> , Hematology <sup>7</sup> , Urinalysis | | X | | | | | | | X |
| 2-hr and 24-hr Urine | | X | | | | | | | X |
| Urine Pregnancy Test <sup>8</sup> | X | X | | X | X | X | X | X | X |
| Vital Signs <sup>9</sup> | X | X | X | X | X | X | X | X | X |
| Height | | X | | | | | | | X |
| Physical Examination | | X | | | | | | | X |
| PHEX mutation analysis | | | | | | | | | |
| Anti-KRN23 antibody (HAHA) <sup>10</sup> | | X | | | | | | | X |
| Serum Phosphorus <sup>11</sup> | | X | X | X | | X | | | X |
| Serum Calcium | | X | X | X | | X | | | X |
| Serum Creatinine | | X | | | | | | | X |
| Serum iPTH | | X | | | | | | | X |
| Serum FGF23 | | X | | | | | | | X |
| Serum 1,25(OH) <sub>2</sub> D | | X | | | | | | | X |
| Bone Biomarkers <sup>12</sup> | | X | | | | | | | X |
| ECHO, ECG | | X | | | | | | | X |

Study Number: UX023-CL203 Statistical Analysis Plan Amendment 1

27 April 2016, Version 1.1



| VISIT TYPE / NUMBER | HH <sup>3</sup> 18 | 19 | HH <sup>3</sup> 20 | НН <sup>3</sup><br>21 | HH <sup>3</sup> 22 | HH <sup>3</sup> 23 | HH <sup>3</sup> 24 | HH <sup>3</sup> 25 | 26 |
|---|---|---|---|---|---|---|---|---|---|
| WEEK <sup>4</sup> | 44 | 48 | 50 | 52 | 56 | 60 | 64 | 68 | 72/<br>EoT <sup>15</sup> |
| WOMAC, BPI, SF36 <sup>13</sup> | | X | | | | | | | X |
| 6MWT, 3MSCT, TUG | | X | | | | | | | X |
| X-Ray <sup>14</sup> | | X | | | | | | | X |
| Interval History | | X | | | | | | | X |
| Prior and Concomitant Medications | X | X | | X | X | X | X | X | X |
| Adverse Events | X | X | | X | X | X | X | X | X |
| Weight | | X | | | | | | | X |
| Drug Administration | X | X | | X | X | X | X | X | |

1,25(OH) <sub>2</sub>D= 1,25-dihydroxy vitamin D; 3MSCT = stair climb test; 6MWT = 6-minute walk test; BL = Baseline; ECG = electrocardiogram; ECHO = echocardiogram; EoT = end of treatment; FGF23 = fibroblast growth factor 23; HAHA = Human Anti-Human Antibody (immunogenicity testing assay); HH = home health; HIV = human immunodeficiency virus; hr = hour; iPTH = intact parathyroid hormone; PHEX = phosphate regulating gene with homology to endopeptidases located on the X chromosome; Scr = Screening; TmP/GFR = the ratio of phosphorus tubule maximum (TmP) to glomerular filtration rate (GFR), or tubular resorption of phosphate; TUG = timed up and go (test)

Screening tests may be spread out over Screening and Baseline assessments, but have to be performed before drug administration. Screening and Baseline visits may be conducted on consecutive days but may be conducted up to 7 days apart.

<sup>2</sup> Baseline Visit tests and assessments may be spread out over 2 consecutive days to accommodate considerable number of assessments.

Home Health (HH) visits may also be conducted at the clinic depending on proximity of the subjects to the investigational site and local availability of home health resources.

The visit window for visits 3 through 25 is  $\pm$  3 days. The visit window for the EoT visit at Week 72 is is  $\pm$  5 days.

Medical history to include review of previous test results for HIV antibody, hepatitis B surface antigen, and/or hepatitis C antibody. Viral testing will not be repeated in this study.

This comprehensive metabolic profile will include the standard Chem-20 serum panel: Na, K, Cl, bicarbonate, blood urea nitrogen (BUN), creatinine and creatinine clearance, glucose, alkaline phosphatase, alanine aminotransferase [ALT], aspartate aminotransferase [AST]), gamma-glutamyl transferase (GGT), lactate dehydrogenase, phosphorus, uric acid, calcium, total protein, albumin, cholesterol and triglycerides, total bilirubin, and indirect bilirubin.

<sup>7</sup> Complete blood count, differential, and platelet count.

For women of childbearing potential only. A serum pregnancy test will be performed in the event of a positive or equivocal urine pregnancy result.



- Vital sign measurements consist of seated systolic/diastolic BP measured in millimeters of mercury (mm Hg), HR (beats per min), respiration rate (breaths per min), and temperature in degrees Celsius (°C). Obtain at the beginning of each visit before any additional assessments are completed.
- If the development of anti-KRN23 antibodies is suspected in a given subject, samples may be obtained at additional time points on a case-by-case basis, if warranted.
- Two serum samples should be collected at clinic visits for serum phosphorus measurements. One sample will be read locally for determination of dosing decision; the other will be sent for analysis by the central laboratory.
- Bone biomarkers will include serum measures of total serum ALP, bone-specific ALP (BALP), CTx, and P1NP.
- Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Brief Pain Inventory (BPI), and SF-36 self-reported patient-reported outcomes (PROs) tools.
- Standard radiographs will be customized by patient and will be repeated every 3 months or until specified lesions are healed.
- Those subjects who terminate the study early will be asked to come back to the clinic for a final assessment. Every reasonable effort should be made to have subjects return to the clinic for the final assessment; however, subjects who are unable to return to the clinic for the final assessment will be given the option of providing blood and urine samples as part of a HH visit.